CLINICAL TRIAL: NCT00350688
Title: Phase II Trial To Evaluate The Potential For Helical Tomotherapy IMRT To Improve Bladder Cancer Chemoradiation
Brief Title: Bladder Cancer Chemoradiation Using Intensity Modulated Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: More advanced treatments superceded study design
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005407-01H; OTT 05-03
Record Dates: First submitted 2006-07-07; First posted 2006-07-11 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Bladder Cancer
Keywords: Bladder,; Cancer,; Chemoradiation,; IMRT,; tomotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Helical tomotherapy IMRT (Other): Helical tomotherapy IMRT
  Interventions: Radiation: Helical tomotherapy IMRT

INTERVENTIONS:
Radiation: Helical tomotherapy IMRT — Helical tomotherapy IMRT

SUMMARY:
While the gold standard of treatment in invasive bladder cancer is surgical removal of the bladder, it is well accepted that a reasonable alternative is an organ preserving approach. Bladder preservation can be achieved in patients with radiotherapy alone or together with concurrent chemotherapy. This clinical trial will assess the potential of intensity modulated radiation therapy (IMRT) delivered using helical tomotherapy to reduce radiation-induced gastrointestinal toxicity and increase the accuracy of bladder cancer irradiation.

DETAILED DESCRIPTION:
Patients opting for bladder conservation in Ottawa are currently treated using intra-arterial cisplatin and concurrent radiotherapy using 3D-Conformal radiotherapy. It has been recently reported that while combination chemotherapy with local therapy (surgery or radiation) does modestly increase survival, greater toxicity results. As a precursor to the integration of gemcitabine in the standard chemotherapy regimen at our centre, the current clinical trial is designed to determine if a novel approach to the delivery of intensity modulated radiotherapy (IMRT), namely Helical Tomotherapy, will decrease the toxicity of standard chemoradiation. Chemoradiation will be administered as follows: 3 courses Intra-Arterial Cisplatin 90mg/m2 every 3 weeks and radical radiation delivered as IMRT for a total dose of 60 Gy in 30 daily fractions of 2 Gy per day M-F starting day 15.

ELIGIBILITY:
Inclusion Criteria:

1. A pathological diagnosis of pure or predominantly transitional cell bladder carcinoma
2. Adequate Hematology and biochemistry parameters
3. Invasive or treatment refractory non-invasive transitional cell bladder carcinoma OR operable patients who prefer bladder preservation OR inoperable patients.
4. No metastases on CT scan of chest

Exclusion Criteria:

1. Patient with contraindication to radical radiotherapy including inflammatory bowel disease or significant irritative bladder symptoms
2. Contraindication to internal iliac arterial catheterization
3. Prior pelvic radiotherapy for other malignancies
4. Prior cytotoxic chemotherapy excepting intravesical agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Acute GI toxicity

SECONDARY OUTCOMES:
Dosimetric evaluation of bowel and pelvic marrow radiation dose, Bladder time organ motion studies, Patterns of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Libni Eapen, MD, Study Director — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario, Canada